CLINICAL TRIAL: NCT04766801
Title: Evaluation of the Efficiency and Complications Associated With the Surgical Treatment of Obesity by Laparoscopic Adjustable Gastric Banding in an Adolescent Population.
Brief Title: Adolescents Bariatric Surgery Cohort Survey
Acronym: BariAdo
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2007-06
Record Dates: First submitted 2020-11-27; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Obesity, Adolescent
Keywords: gastric banding; complications; weight loss
MeSH Terms: conditions — Obesity, Morbid; Pediatric Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic adjustable gastric banding — Weight-loss surgery, with the use of gastric banding

SUMMARY:
Obesity affects 3%-4% of the pediatric population and leads to cardiac mortality during adult life. Bariatric surgery is the best treatment for weight loss and preventing obesity associated comorbidities in adults, but its applications and safety are yet to be defined for adolescents.

DETAILED DESCRIPTION:
Since 2008, in France, certain university hospitals have been eligible to perform bariatric surgery for adolescents. It was therfore possible to define its feasibility, potential complications and specific indications.

This led to recommandations published by Health Authorities (HAS) in 2016. However, it seems imperative to continue monitoring these patients in order to improve their management, especially as the use of these surgical techniques becomes increasingly widespread.

The Angers University Hospital is one of the leading hospitals when it comes bariatric surgery for adolescents through its use of gastric bands.

The aim of this protocol is to update data on how effective this surgery is on weight loss and obesity-associated comorbidities, and to monitor medical, psychological and surgical complications associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14-20 years of age and asking for bariatric surgery
* BMI >= 40 Kg.m-2 or >= 35 Kg.m-2 with major obesity-related comorbidities (hypertension, diabetes, sleep apnea, etc...)

Exclusion Criteria:

* An unstable psychiatric disorder
* Bariatric surgery anesthesic contraindications
* Having not completed a minimum of six months of the pre operative program
* Lack of consent from the patient or the patient's relatives.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients treated in our hospital for morbid obesity (BMI >= 35 Kg.M-2) through different programs with lifestyle and nutritional interventions and, for those who requested it, the possibility of bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of weight parameters at 2 years compared to preoperative baseline | 2 years
  Evaluation of weight loss by weight (Kg), body mass index (BMI, Kg.m-2) and excess body weight (EBWL, %) changes

SECONDARY OUTCOMES:
Changes of insulin resistance at 2 years | 2 years
  Evaluation of insulin resistance by measure of the HOMA index
Evaluation of dyslipidemia | 2 years
  Evaluation of lipid profile (cholesterol, triglycerides)
Evaluation of liver steatosis | 2 years
  Evaluation of liver steatosis and NAFLD on US exam and liver elastometry
Resolution of comorbidities associated with obesity | 2 years
  Clinical evaluation of the presence/absence of hypertension, sleep apnea, orthopedic disorders and polycystic ovary at two years, compared to Baseline characteristics
Monitoring of psychiatric profile | 2 years
  Clinical evaluation of the presence/absence of psychiatric disorders such as binge eating, depression, etc...
Evaluation of quality of life | 2 years
  Evaluation of obesity-related QOL by the use of the PedsQL scale
Evaluation of cosmetic satisfaction | 12 months postoperative
  Evaluation of the patient's level of satisfaction with regards to their surgical scar using the POSAS scale
Surgical complications | 2 years
  Monitoring of the occurrence of surgical complications and their severity thanks to the Clavien-Dindo scale at each medical consultation

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Schmitt, MD-PhD, Principal Investigator — University Hospital of Angers
Locations (1):
- University Hospital of Angers, Angers, Maine Et Loire, France